CLINICAL TRIAL: NCT05810116
Title: Effect of Palmitoylethanolamide (PEA) Compared to a Placebo on Acute Menstrual Pain in an Adult Population - a Double-blind, Crossover, Randomised Controlled Trial.
Brief Title: Effectiveness of PEA Compared to Placebo on Acute Menstrual Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEAMPS-23
Record Dates: First submitted 2023-03-27; First posted 2023-04-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-03

CONDITIONS: Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levagen+ (Active Comparator): PEA in capsule form - 1 capsule with water upon pain onset, followed by another capsule with water after 2 hours if pain persists.
  Interventions: Drug: Levagen+
- Microcrystalline cellulose (Placebo Comparator): PEA in capsule form - 1 capsule with water upon pain onset, followed by another capsule with water after 2 hours if pain persists.
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: Levagen+ — Daily dose of 1-2 capsules (1 capsule containing 350mg Levagen+ equivalent to 300mg PEA)
  Arms: Levagen+
Drug: Microcrystalline cellulose — Daily dose of 1-2 capsules (1 capsule containing 350mg)
  Arms: Microcrystalline cellulose

SUMMARY:
This is a double blind, randomised, placebo-controlled trial to evaluate orally-dosed Palmitoylethanolamide (PEA) compared to placebo on menstrual pain in otherwise healthy participants 18 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Women who experience mild to moderate menstruating pain
* Aged 18 years or over
* History of over the counter (OTC) analgesic use for the treatment of menstrual pain
* Self-reported history of menstrual cramp pain occurring during four of the past six menstrual cycles.
* Typically requires at least one dose of an OTC analgesic medication such as naproxen, aspirin, ibuprofen or acetaminophen taken on at least 1 day of menstrual cycle for the treatment of mild to moderate menstrual cramp, and normally experiences pain relief from these medications.
* Otherwise healthy
* Able to provide informed consent
* Regular menstrual cycle (28 days ± 7 days) and period
* Agree not to participate in any other clinical trial while enrolled in this trial

Exclusion Criteria:

* Secondary cause for dysmenorrhea (i.e. endometriosis, adenomyosis, uterine fibroids or infection)
* Any bleeding disorders, recent surgery or concurrent blood thinning treatment
* Unstable or serious illness (e.g., kidney, liver, GIT, heart conditions, diabetes, thyroid gland function, lung conditions, chronic asthma, diagnosed psychological or mood disorder) (1)
* Current malignancy (excluding BCC) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy
* Pregnant or lactating women
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic or hypersensitive to any of the ingredients in active or placebo formula
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participated in any other clinical trial during the past 1 month

  1. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Change in acute menstrual pain severity, analgesic effect via Numeric Rating Scale (NRS) | 4 menstrual pain events over a maximum of 16 weeks
  Reduction in acute menstrual pain severity, analgesic effect via Numeric Rating Scale (NRS) a pain assessment tool commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". The higher the score the worse the pain.

SECONDARY OUTCOMES:
Change in categorical pain levels via categorical pain relief scale | 4 menstrual pain events over a maximum of 16 weeks
  Reduction in categorical pain levels via categorical pain relief scale (better, much better, no change, worse, much worse)
Effectiveness of the Treatment via Global Satisfaction scale of the Treatment Satisfaction Questionnaire for Medication (TSQM) | 4 menstrual pain events over a maximum of 16 weeks
  Effectiveness of the Treatment via Global Satisfaction scale of the Treatment Satisfaction Questionnaire for Medication (TSQM). To assess the overall level of satisfaction or dissatisfaction with medication patients are taking. Higher scores indicate higher satisfaction.
Change in rescue medication use via self-report | 4 menstrual pain events over a maximum of 16 weeks
  Change in rescue medication use via self-report
Safety of Use | From enrolment and until 4 menstrual pain events are recorded - a maximum of 16 weeks
  Safety via Adverse Event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, New Farm, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared